CLINICAL TRIAL: NCT00237588
Title: Glucose Optimisation With Angiotensin II Antagonist Losartan in Patients With Hypertension and Other Risk Factors for Metabolic Syndrome (GOAAL)
Brief Title: Glucose Optimisation With Angiotensin II Antagonist Losartan (GOAAL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 308-1
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2005-10

CONDITIONS: Hypertension
Keywords: Angiotensin II Type I Receptor Blockers; Amlodipine; Calcium Channel Blockers; Diabetes Mellitus; Hypertension; Insulin Resistance; Losartan
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Insulin Resistance | interventions — Amlodipine; Losartan

INTERVENTIONS:
Drug: Amlodipine 10 mg or Losartan 100 mg + Amlodipine 5 mg

SUMMARY:
To determine if angiotensin-II AT-1 receptor blockade(ARB) may improve insulin sensitivity assessed by the hyperinsulinaemic isoglycaemic glucose clamp, more than CCB therapy at a comparable dose with regards to the blood pressure-lowering effect.

DETAILED DESCRIPTION:
Patients with hypertension have an increased prevalence of insulin resistance and an increased risk of developing diabetes mellitus with ageing. Different antihypertensive regimens have varying effects on glucose metabolism and the development of diabetes mellitus. In a double-blind,randomized cross-over study we aim to compare the metabolic effects of 10 mg amlodipine and 100 mg losartan + 5 mg amlodipine in patients with hypertension and other risk factors for the metabolic syndrome.

After a 4-week open label amlodipine 5 mg run-in period, all hypertensive patient will be randomized to additional treatment with either amlodipine 5 mg or losartan 100 mg for 8 weeks. At the end of this 8-week treatment-period we will do a physical examination, laboratory-tests, hyperinsulinaemic isoglycaemic glucose clamp, heart rate variability and baroreflex sensitivity measurements. Following this is a 4-week wash-out phase where the subjects continue open label 5 mg amlodipine, before crossed over to the opposite treatment regimen for another 8 week before the final examination.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension with diastolic blood pressure 95-110 mmHg and systolic blood pressure < 180 mmHg
* Previously untreated hypertension or treated with monotherapy (but not with ACE-inhibitors or Angiotensin II-receptor blockers)
* Impaired glucose tolerance or impaired fasting glucose (fasting plasma glucose; 6.1-7.0 mmol/l (110-126 mg/dl)
* Age over 18
* Informed consent
* Any one of these: Microalbuminuria (urin excretion >20 microg/min), dyslipidemia (HDL-cholesterol <0.9 mmol/l(35 mg/dl), Triglycerides > 1.7 mmol/l (150 mg/dl), waist to hip-ratio >0.9 in men and >0.85 in women, BMI >28 kg/m2.

Exclusion Criteria:

* Previous or current use of ACE-inhibitors or Angiotensin II-receptor blockers
* Previous or current antidiabetic medications
* "Brittle" pre-diabetes where the investigator anticipates pharmacological treatment within next 6 months
* Hypertensive patients where the investigator anticipates polytherapy within next 6 months
* Female patient who is pregnant or nursing or planning pregnancy within the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-12; Study Completion 2005-07

PRIMARY OUTCOMES:
Insulin sensitivity assessed with hyperinsulinaemic isoglycaemic glucose clamp(GDR)

SECONDARY OUTCOMES:
Fasting serum glucose
Fasting serum insulin
HOMA-IR
C-peptide
High sensitivity C-reactive protein
Lipids (Triglycerides, Total-cholesterolHDL-cholesterol, LDL-cholesterol)
Adipocytokines etc.(Adiponectin, leptin, resistin, TNF-a, PAI-1 activity, ghrelin)
Serum uric acid
Catecholamines
Baroreflex sensitivitiy
Heart rate variability
Microalbuminuria

CONTACTS AND LOCATIONS:
Overall Officials: Sverre E Kjeldsen, MD, PhD, Study Director — Ullevaal University Hospital
Locations (1):
- Cardiovascular and Renal Research Center/ Department of Cardiology, Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Result] Aksnes TA, Reims HM, Guptha S, Moan A, Os I, Kjeldsen SE. Improved insulin sensitivity with the angiotensin II-receptor blocker losartan in patients with hypertension and other cardiovascular risk factors. J Hum Hypertens. 2006 Nov;20(11):860-6. doi: 10.1038/sj.jhh.1002087. Epub 2006 Sep 21. PMID 16988754
- See also: Homepage for Cardiovascular and Renal Research Center, Ullevaal University Hospital, Oslo, Norway — http://www.cvr.no